CLINICAL TRIAL: NCT04179084
Title: Phase II Study to Evaluate the Efficacy and Safety of Fruquintinib Plus Sintilimab as Third-line Therapy for Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fruquintinib
Record Dates: First submitted 2019-11-07; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Metastasis Colorectal Cancer
MeSH Terms: interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fruquintinib + Sintilimab (Experimental)
  Interventions: Drug: fruquintinib; Drug: Sintilimab

INTERVENTIONS:
Drug: fruquintinib — 5mg qd, 2weeks on, 1week off
Drug: Sintilimab — 200mg q3w

SUMMARY:
This study is a single center, investigator initiated phase II clinical study to evaluate the efficacy and safety of fruquintinib plus Sintilimab as third-line therapy for colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

- Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.

Subjects with metastatic colorectal cancer(CRC) (Stage IV). Subjects must have failed at least two lines of prior treatment. Progression during or within 3 months following the last administration of approved standard therapies which must include a fluoropyrimidine, oxaliplatin and irinotecan.

Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy.

Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible.

Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study.

Subjects may have received prior treatment with Avastin (bevacizumab) and/or Erbitux (cetuximab)/Vectibix (panitumumab) (if KRAS WT) Metastatic CRC subjects must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1.

Eastern Cooperative Oncology Group (ECOG) Performance Status of 1. Life expectancy of at least 12 weeks. Adequate bone marrow, liver and renal function as assessed by the laboratory required by protocol.

Exclusion Criteria:

- Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody, anti-cytotoxic T lymphocyte-associated antigen 4 (cytotoxic T-lymphocyte-associated Protein 4, CTLA-4) antibody or other drug/antibody that acts on T cell costimulation or checkpoint pathways.

Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].

Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization.

Cardiological disease including Congestive heart failure, Unstable angina, Myocardial infarction, Cardiac arrhythmias requiring anti-arrhythmic therapy.

Uncontrolled hypertension. (Systolic blood pressure 150 mmHg or diastolic pressure 90 mmHg despite optimal medical management).

Pleural effusion or ascites that causes respiratory compromise. Arterial or venous thrombotic or embolic events. Any history of or currently known brain metastases. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.

Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 4 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1year
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR).

SECONDARY OUTCOMES:
Overall Survival (OS) | 1year
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
Progression-free survival (PFS) | 1year
  The PFS is defined as the time from the start of treatment to the date of first documented PD or death as a result of any cause, whichever occurred first. When a patient was alive and without progression, PFS was censored at the date of the last disease assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- China PLAGH, Beijing, China

IPD SHARING:
Plan to Share IPD: No